CLINICAL TRIAL: NCT03060057
Title: Prospective Post Approval Clinical Follow-Up Study of the Commercially Available U2 Knee™ System - "U-Propel Study"
Acronym: U-Propel
Status: Active, not recruiting | Type: Observational
Sponsor: United Orthopedic Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 03-2017
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: U2 Knee™ System — The United U2 Knee™ System consists of several components and for this clinical evaluation it includes the (1) Femoral Component, (2) Tibial Insert, 3) Tibial Baseplate, and the 4) Patella.

SUMMARY:
The purpose of this study is to evaluate both short and long term clinical performance and safety of the commercially available U2 Knee™ System.

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-center, post-approval study designed to evaluate the short and long term clinical performance and safety in subjects receiving primary total knee arthroplasty (TKA) with the U2 Knee™ System. The study will enroll up to 200 subjects with scheduled pre-discharge, 6-week, 3- and 6-month and up to 5-year annual follow-up visits. Study outcomes will be analyzed and published when 1.) all enrolled and implanted subjects complete their 6-week follow up, 2.) all implanted subjects complete their 2-year follow up, 3.) at the conclusion of the study.

The study will follow GCP guidelines and will be registered on clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 75 years of age
2. Subject is indicated for a unilateral total knee arthroplasty (TKA) based on the approved labeling of the device
3. Subject has no history of previous prosthetic replacement device or orthopedic surgeries on the operative knee
4. Subject is willing and able to provide informed consent to participate in the study;
5. Subject is willing and able to understand the purpose of the study, his/her role, and is available to return to the clinic/hospital for all required follow-up visits;

Exclusion Criteria:

* Subjects will be excluded if, in the opinion of the Investigator, the subject does not qualify based on approved labeling requirements or Subject Inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The U2 Knee™ System is intended for use in subjects who require primary total knee arthroplasty for reduction or relief of pain and/or improved knee function.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 2 Years
  Device Survivorship defined as no revision of removal of any parts of the system

SECONDARY OUTCOMES:
Change in Knee Society Score (KSS) Over Time | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, 5 years
  This endpoint is defined as differences in both pain and functional parameters measured at current and pre-discharge visits
Change in EQ-5D Over Time | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, 5 years
  This endpoint is defined as differences in scores related to the EQ-5D questionnaire and the EQ-VAS measured at current and pre-discharge visits.
Change in EQ-5D VAS Over Time | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, 5 years
  This endpoint is defined as differences in scores related to the EQ-5D VAS questionnaire and the EQ-VAS measured at current and pre-discharge visits.
Change in KOOS, JR. Over Time | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 3 years, 4 years, 5 years
  This endpoint is defined as difference in the KOOS, Jr interval score measured at current and pre-discharge visits.
Radiographic Analysis | 24 months, 5 years
  This endpoint is defined as incidence rate of new radiographic failures at each follow-up visit.
Operative characteristics | Operative
  Descriptive statistics in operative characteristics will be reported as secondary endpoints to evaluate operative success
Subject Satisfaction Survey | 6 weeks, 3 months, 6 months, 12 months, 2 Years, 3 Years, 4 Years and 5 Years.
  Subject satisfaction with their knee surgery.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Coastal Orthopedics, Bradenton, Florida
  - Jacksonville Orthopaedic Institute, Jacksonville, Florida
  - Orthopedic Center of Vero Beach, Vero Beach, Florida
  - Rubin Institute for Advanced Orthopedics, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided